CLINICAL TRIAL: NCT03634371
Title: Bioequivalence Study of Levothyroxine Sodium Tablets 150 mcg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tecnoquimicas (Industry)
Responsible Party: Principal Investigator, Mauricio Vargas, Biopharmaceutical Studies Director, Tecnoquimicas
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Versión 3- BIO 096
Record Dates: First submitted 2018-08-12; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formulation of Levothyroxine (Experimental): Levothyroxine sodium tablets 150 mcg Single dose of 600 mcg administered in dosing period 1 or 2
  Interventions: Drug: Drug Levothyroxine 150 mcg
- Reference formulation of Levothyroxine (Active Comparator): Eutirox 150 mcg Single dose of 600 mcg administered in dosing period 1 or 2
  Interventions: Drug: Drug Eutirox 150 mcg

INTERVENTIONS:
Drug: Drug Levothyroxine 150 mcg — Administration of a 600 mcg levothyroxine dose
  Arms: Test Formulation of Levothyroxine
Drug: Drug Eutirox 150 mcg — Administration of a 600 mcg levothyroxine dose
  Arms: Reference formulation of Levothyroxine

SUMMARY:
The objective of this study is to establish the bioequivalence of two levothyroxine formulations through the estimation of T4 levels in serum samples after baseline correction, according to Food and Drugs Administration (FDA), World Health Organization (WHO) and Colombian National Vigilance Institute for Drugs and Food (INVIMA) guidelines.

DETAILED DESCRIPTION:
Levothyroxine (T4) is used to treat patients with hypothyroidism and may often result in lifelong therapy. Its physiologically active metabolite is tri-iodothyronine (T3). Levothyroxine is also endogenously produced in the body. Since small changes in levothyroxine administration (e.g. change in brand or formulation) can cause significant changes in serum thyroid stimulating hormone (TSH) concentrations, precise and accurate TSH control is critical to avoid potential adverse iatrogenic effects. Tecnoquimicas modified its Levothyroxine tablets formulation in order to comply with new pharmacopeical specifications. It will then evaluate the impact on drug product performance based on pharmacokinetic (PK) measures of total serum T4 and total serum T3 of the new formulation of levothyroxine (Test formulation) relative to the reference formulation from Merck (Reference formulation)

This will be a single-center, open-label, two-period, two-treatment, two-sequence, randomized, single-dose, crossover study. 80 healthy adults will be randomized to receive a single dose (4 x 150 mcg tablets = 600 mcg) of the test formulation of levothyroxine and reference formulation of levothyroxine separately in each treatment period. There will be two treatment sequences (AB, BA) and a 42 day washout between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women from 18 to 50 years old
* Diagnosed as healthy after a clinical examination
* BMI from 18 to 30 kg/m2
* Not smoking for at least 3 months
* To sign the informed consent
* Not having participated in a similar study for at least 4 months

Exclusion Criteria:

* Renal, cardiac immunological, dermatological, endocrine, gastrointestinal, neurological or psychiatric condition
* Hematologic disorders, specially anemia and polycythemia
* Permanent or temporal pharmacological therapy, prescribed or not
* Smoking for the last 3 months
* Alcohol drinker more than once a week
* Drug abuse
* Drug hypersensitivity
* Angioedema or anaphylaxis history
* Pregnancy or breast-feeding
* HIV o Hepatitis B diagnosed
* Blood donor in the past 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-10-06 (Estimated); Study Completion 2018-10-06 (Estimated)

PRIMARY OUTCOMES:
(AUC) Area Under the Curve 0-48 for T4 | From 0 to 48 hours
  -0.5, -0.25, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours
Cmax for T4 | From 0 to 48 hours
  -0.5, -0.25, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours

SECONDARY OUTCOMES:
AUC 0-48 for T3 | From 0 to 48 hours
  -0.5, -0.25, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours
Cmax for T3 | From 0 to 48 hours
Tmax | From 0 to 48 hours
  -0.5, -0.25, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours
Kel | From 0 to 48 hours
  -0.5, -0.25, 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de la Sabana, Chía, Colombia

IPD SHARING:
Plan to Share IPD: No